CLINICAL TRIAL: NCT00717847
Title: A Study of Serum Protein Profiling in Patients With Non-Small Cell Lung Cancer Treated With Gefitinib or Erlotinib
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Other Study IDs: NS01/19/05
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- 1: Any patient with NSCLC receiving erlotinib or gefitinib
- 2: Patients with unexpected and/or severe treatment related toxicity whilst receiving EGFR TKI.

SUMMARY:
We hypothesize that Epidermal growth factor receptor tyrosine kinase inhibitors modulate tumor changes that may be reflected in the alteration of serum proteins.

Study objectives are:

* To establish serum proteomic changes in patients with non-small cell lung cancer (NSCLC) receiving erlotinib or gefitinib.
* To identify a serum protein profile that predicts erlotinib or gefitinib sensitivity or resistance in NSCLC patients with and without EGFR mutations.
* To study the toxicity of erlotinib or gefitinib by correlating clinical toxicity with serum protein profile.

DETAILED DESCRIPTION:
Background:

Although some success has been achieved in identifying Epidermal growth factor receptor (EGFR) mutations as a molecular predictive marker of response in patients with non-small cell lung cancer (NSCLC), this strategy is likely only to be limited as not all responding patients have a mutation in their tumor and conversely, not all patients with a mutation were responders. Furthermore, as the development of resistance to EGFR tyrosine kinase inhibitors (TKI) such as gefitinib, erlotinib is inevitable and poses a major clinical problem due to limited therapeutic options, the identification of a molecular profile that could predict sensitivity to erlotinib or gefitinib is warranted.

Hypothesis:

Using serum as an easily accessible biological fluid, we hypothesize that EGFR TKIs modulate tumor changes that may be reflected in the alteration of serum proteins.

Objectives:

* To establish the serum proteomic changes in NSCLC patients receiving erlotinib or gefitinib.
* To identify a serum protein profile that predicts erlotinib or gefitinib sensitivity or resistance in NSCLC patients with and without EGFR mutations.
* To study the toxicity of erlotinib or gefitinib by correlating clinical toxicity with serum protein profile.

Significance:

An extensive profiling of the molecular circuitry affected by EGFR TKIs would be helpful in understanding the response and side effects of patients with NSCLC treated with erlotinib or gefitinib and could guide therapy and thus improve patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with NSCLC receiving erlotinib or gefitinib.
* Patients with unexpected and/or severe treatment related toxicity whilst receiving EGFR TKI.
* Age ≥ 18 years
* Written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with NSCLC receiving erlotinib or gefitinib. Patients with unexpected and/or severe treatment related toxicity whilst receiving EGFR TKI.
Sampling Method: Probability Sample
Dates: Start 2006-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ross Andrew Soo, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore